CLINICAL TRIAL: NCT05115006
Title: Adjuvant Melanoma Stakeholder Treatment Preference Study
Brief Title: A Study of Adjuvant Melanoma Stakeholder Treatment Preferences
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8YR
Record Dates: First submitted 2021-10-28; First posted 2021-11-10 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Melanoma
Keywords: Melanoma; Discrete choice experiment; Resected melanoma; Adjuvant treatment; Patient preference
MeSH Terms: conditions — Melanoma; Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Cohort 1: Participants diagnosed with stage II and stage III melanoma who have undergone surgery

SUMMARY:
The purpose of this study is to understand the trade-offs that participants with surgically treated melanoma would be willing to make among key features and outcomes of adjuvant anti-cancer treatments or no adjuvant treatment / observation.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported medical diagnosis of stage II or stage III melanoma
* Have been resected (had surgery) for their melanoma within 12 months prior to study participation

Exclusion Criteria:

* Self-reported stage IIa
* Self-reported recurrence of melanoma after surgery

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is to include 350 adult participants from the US, Australia, UK, Germany, France, Spain, and Italy who self-report to have stage IIb, IIc, or III melanoma and who have had surgery for melanoma within 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Preference weights or utilities (a measure of relative preference; on a continuous variable scale) for each treatment attribute level based on responses to the Discrete Choice Experiment (DCE) choice tasks | At Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Melbourne, Victoria, Australia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm